CLINICAL TRIAL: NCT03796806
Title: Methods Validation Assessment for Study of Inflammatory Skin Disease
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Julia S. Lehman, Professor of Dermatology and Laboratory Medicine and Pathology, Mayo Clinic
Other Study IDs: 18-002404
Record Dates: First submitted 2018-10-22; First posted 2019-01-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Lichen Planus
Keywords: lichen planus; proteomics; xenograft model for lichen planus
MeSH Terms: conditions — Lichen Planus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Assess validity of methods involved in molecular studies of the skin in inflammatory skin disease
2. Assess feasibility of methods for grafting fresh human skin (normal and diseased with inflammatory skin disease) onto an established xenograft murine model.

DETAILED DESCRIPTION:
The use of fixed tissue specimens for research studies is attractive, because a large number of relevant specimens can be collected quickly from tissue registry. There is a current lack of knowledge regarding to what extent formalin fixation alters the identification of proteins in the skin with inflammatory dermatoses. This information would be important to assess when determining the limitations (or potentially lack thereof) of using fixed specimens in research.

Collaborators have successfully developed a murine model that can accept human skin xenografts. While those investigators have successfully demonstrated transplantation of healthy skin onto mice, it is unknown whether skin affected by inflammatory disease can be transplanted and, if so, whether the inflammatory skin disease remains, whether it spreads to involve host skin, or whether it resolves. Determining feasibility of transplanting inflamed human skin using this model, as well as observing the course of this inflammation, are the next steps in advancing this potentially invaluable research modality.

ELIGIBILITY:
Inclusion Criteria:

- Adults >18 years with active cutaneous lichen planus with capacity to consent.

Exclusion Criteria:

* Concurrent skin infection
* Wound healing disturbances
* Patients on systemic immunosuppressive medications.
* Lidocaine allergy
* Platelets <10,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinic patients with active lichen planus and residing within a 50-mile radius of Mayo Clinic-Rochester.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Comparative analysis of proteomes on fresh versus formalin-fixed-paraffin-embedded tissue. | 8 months
  Identification and quantification of proteins as obtained by liquid chromatography-mass spectrometry methods using fresh and formalin-fixed-paraffin-embedded tissue. Mass spectrometry data will be matched against a composite protein sequence database using the MyriMatch search engine and IDPicker will filter protein identification at 2% false discovery rate. QuasiTel software will process the spectral count data for the identification of differentially expressed proteins.
Viability of human inflammatory skin (lichen planus) graft in a xenograft murine model | 8 months
  Viability of diseased human graft into an established murine xenograft model by visual inspection and microscopic analysis.
Evaluation of inflammation around human inflammatory skin graft (lichen planus) and elsewhere in a established xenograft murine model | 8 months
  Assessment of inflammation around graft and elsewhere in the host by visual inspection and microscopic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Julia S Lehman, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials